CLINICAL TRIAL: NCT00590174
Title: Evaluation of the Long-term Safety After Zotarolimus-Eluting Stent, Sirolimus-Eluting Stent, or PacliTaxel-Eluting Stent Implantation for Coronary Lesions - Late Coronary Arterial Thrombotic Events
Brief Title: Clopidogrel Use and Long-term Safety After Drug-Eluting Stents Implantation
Acronym: ZEST-LATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20070043
Record Dates: First submitted 2007-12-31; First posted 2008-01-10 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Coronary Artery Disease
Keywords: stent; antiplatelet therapy
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Experimental): Aspirin monotherapy (stopping clopidogrel at 1 year after DES)
  Interventions: Drug: Aspirin
- Aspirin,Clopidogrel (Active Comparator): Aspirin,Clopidogrel Dual antiplatelet therapy (continue aspirin and clopidogrel 1year after DES)
  Interventions: Drug: Aspirin,Clopidogrel

INTERVENTIONS:
Drug: Aspirin — stopping clopidogrel at 1 year after DES implantation
  Other Names: Aspirin monotherapy
  Arms: Aspirin
Drug: Aspirin,Clopidogrel — continue aspirin and clopidogrel 1year after DES
  Other Names: Aspirin,Clopidogrel Dual antiplatelet therapy
  Arms: Aspirin,Clopidogrel

SUMMARY:
The purpose of ZEST-LATE (Evaluation of the Long-term Safety After Zotarolimus-Eluting Stent, Sirolimus-Eluting Stent, or PacliTaxel-Eluting Stent Implantation for Coronary Lesions - Late Coronary Arterial Thrombotic Events) trial is to assess the relationship between long-term clopidogrel use beyond 1 year and long-term rates of death or MI after DES implantation and to estimate the duration of dual antiplatelet therapy for preventing the late thrombotic events.

DETAILED DESCRIPTION:
Prospective, two arms, open-labeled, randomized multi-center trial of approximately 2,000 patients enrolled at 19 centers in Korea. Among all patients enrolled in the ZEST (Comparison of the Efficacy of Zotarolimus-Eluting Stent versus Sirolimus-Eluting Stent versus PacliTaxel-Eluting Stent for Coronary Lesions) trial, event-free patients who survived the first 12 months without nonfatal MI or repeat revascularization will be randomized to discontinue clopidogrel therapy at 12 months after DES implantation. All patients will be followed for another 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Among the participants in the ZEST trial, event-free patients who survived the first 12 months without nonfatal MI or repeat revascularization
2. The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

1. Contraindication to antiplatelet therapy
2. Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
3. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
4. Bleeding diathesis
5. Recent stroke within 6-months
6. Concurrent organ damage (creatinine level > 2.0mg/dL or AST and ALT > 3 times upper normal reference values)
7. Patients with left main stem stenosis (>50% by visual estimate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1175 (Actual)
Dates: Start 2007-10; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Composite of death or myocardial infarction | at 12 months after randomization (at 24 months after ZEST enrollment)

SECONDARY OUTCOMES:
All Death | at 12 months after randomization
Cardiac death | at 12 months after randomization
Myocardial infarction | at 12 months after randomization
Stroke | at 12 months after randomization
Target vessel revascularization (all and ischemia-driven) | at 12 months after randomization
Target lesion revascularization (all and ischemia-driven) | at 12 months after randomization
Stent thrombosis for the patients | at 12 months after randomization
Bleeding event | at 12 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Department of Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (20):
- South Korea (20):
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Asan Medical Center, Gangneung
  - Chonnam National University Hospital, Gwangju
  - NHIC Ilsan Hospital, Ilsan
  - Chonbuk National University Hospital, Jeonju
  - Pusan Natioanal University Hospital, Pusan
  - Hallym University Sacred Heart Hospital,, Pyeongchon
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - St.Mary's Catholic Medical Center, Seoul
  - Yonsei University Medical Center, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hospital, Ulsan
  - Yonsei University Wonju Christian Hospital, Wŏnju

REFERENCES:
- [Derived] Park SJ, Park DW, Kim YH, Kang SJ, Lee SW, Lee CW, Han KH, Park SW, Yun SC, Lee SG, Rha SW, Seong IW, Jeong MH, Hur SH, Lee NH, Yoon J, Yang JY, Lee BK, Choi YJ, Chung WS, Lim DS, Cheong SS, Kim KS, Chae JK, Nah DY, Jeon DS, Seung KB, Jang JS, Park HS, Lee K. Duration of dual antiplatelet therapy after implantation of drug-eluting stents. N Engl J Med. 2010 Apr 15;362(15):1374-82. doi: 10.1056/NEJMoa1001266. Epub 2010 Mar 15. PMID 20231231